CLINICAL TRIAL: NCT06981286
Title: Oral Health Parameter-Based Diabetes Type 2 Indication Using Machine Learning in Older Individuals With Mild Cognitive Impairment
Brief Title: Oral Health Parameter-Based Diabetes Type 2 Indication Using Machine Learning
Acronym: JFG
Status: Not yet recruiting | Type: Observational
Sponsor: Blekinge Institute of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: DT2 prediction
Record Dates: First submitted 2025-04-07; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes
Keywords: Oral Health; Machine Learning; Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- T2D: Older individuals with Diabetes type 2
  Interventions: Other: A dataset comprising participants withT2D will be used to evaluate the classification performance of various machine learning techniques.
- Group/Cohort Description: Older individuals without Diabetes type 2

INTERVENTIONS:
Other: A dataset comprising participants withT2D will be used to evaluate the classification performance of various machine learning techniques. — A dataset comprising participants with T2D will be used to evaluate the classification performance of various machine-learning techniques.
  Groups: T2D

SUMMARY:
This study aims to explore the potential of using machine learning (ML) algorithms to predict Diabetes type2, based on oral health and demographic data. The objective is to evaluate the effectiveness of various ML models and identify the most relevant oral health indicators for predicting type 2 diabetes in individuals with mild cognitive impairment aged 60 and above.

DETAILED DESCRIPTION:
This cross-sectional study utilizes oral health and demographic data from the Swedish National Study on Aging and Care (SNAC-B). Participants aged 60 years or older with Mild Cognitive Impairment will be included in the analysis. The data will be used to develop and evaluate machine learning models for predicting type 2 diabetes.

Objectives:

1. Primary Objective: To assess the potential of oral health parameters for binary classification of type 2 diabetes or not.
2. Secondary Objective: To identify the most influential oral health parameters contributing to type 2 diabetes predictions.
3. Tertiary Objective: To compare the performance of Random Forest (RF), Support Vector Machine (SVM), and CatBoost (CB) classifiers in predicting type 2 diabetes using oral health data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years or older.
* Participants with recorded oral health parameters with or without Diabetes type2

Exclusion Criteria:

• Individuals with Diabetes type1

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Data collected from the Swedish National Study on Aging and Care (SNAC-B) will be analyzed. Participants aged 60 years or older will be included in the analysis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Detection perfomance | 12 months
  Description: The study measures the classification performance of Machine Learning classifier. Performance metrics, Accuracy, precision, recall, F1-Score and confusion matrix will be used for the evaluation. The examination of the most important features relied on SHAP summary plots, providing visualizations of the influence of parameter groups on the output, organized by their importance. This importance is based on SHAP values, offering insights into features' effects on the ML model's decision-making process

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Health, Blekinge Institute of Technology, Karlskrona, Sweden

IPD SHARING:
Plan to Share IPD: No
Participant data can not be shared due to the GDPR.